CLINICAL TRIAL: NCT07328243
Title: Efficacy of Irreversible Electroporation Ablation for Postoperative Recurrent or Metastatic Cervical Lymph Node Disease in Thyroid Cancer: A Prospective, Multicenter, Single-Arm, Exploratory Clinical Trial
Brief Title: Irreversible Electroporation for Recurrent or Metastatic Cervical Lymph Node Metastases From Thyroid Cancer: A Prospective Multicenter Single-Arm Study
Acronym: IRE-TCLN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tian'an Jiang (Other)
Responsible Party: Sponsor-Investigator, Tian'an Jiang, The First Affiliated Hospital, Zhejiang University School of Medicine, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20250178C-R1; MR-33-25-085936 (Registry Identifier: Medical Research Registration and Filing Information System (China))
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Thyroid Cancer Patients; Lymph Node Metastasis
MeSH Terms: conditions — Lymphatic Metastasis | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IRE Ablation (Experimental): Participants with postoperative recurrent or metastatic cervical lymph node disease from thyroid cancer will undergo ultrasound-guided IRE ablation on Day 0. Imaging re-assessment will be performed at Day 30 (±7 days). If residual enhancement suggests incomplete ablation, one salvage IRE ablation may be performed within 14 days per protocol.
  Interventions: Device: Irreversible Electroporation (IRE) Ablation

INTERVENTIONS:
Device: Irreversible Electroporation (IRE) Ablation — Ultrasound-guided IRE ablation of target cervical lymph node(s). A salvage IRE ablation may be performed within 14 days after the Day 30 (±7 days) imaging assessment if incomplete ablation is suspected.

SUMMARY:
This is a single-arm, open-label, multicenter, exploratory clinical trial designed to systematically evaluate the efficacy, safety, and patient benefit of ultrasound-guided irreversible electroporation (IRE) ablation for recurrent or metastatic cervical lymph node disease in patients with thyroid cancer after prior curative thyroid surgery and neck dissection. A total of 85 participants will be enrolled.

After providing written informed consent, participants will enter a screening period of up to 28 days. During screening, baseline imaging of target lymph nodes will be performed (contrast-enhanced ultrasound or computed tomography), and patient-reported and clinician-reported assessments will be completed, including quality of life, pain, neck appearance, and, when applicable, voice-related outcomes. Laboratory testing and immunology samples will also be collected.

Eligible participants will undergo the first IRE ablation on Day 0 under ultrasound guidance. Acute pain will be assessed using the Numeric Rating Scale (NRS) at 0, 4, 8, 24, 48, and 72 hours after the procedure, and all adverse events and device deficiencies will be recorded. The first imaging re-assessment will be performed at Day 30 (±7 days). If residual enhancement suggests incomplete ablation, one salvage IRE ablation may be performed within 14 days. After confirmation of no need for salvage ablation or after completion of salvage ablation, participants will enter follow-up.

Follow-up visits will occur every 3 months starting from Month 3 after the first (or salvage) ablation and will continue until 24 months or until imaging progression, withdrawal, death, or loss to follow-up, whichever occurs first. Imaging assessments will be performed at each follow-up visit. At 12 months, the volume reduction rate (VRR), complete disappearance rate, and recurrence rate of treated lymph nodes will be assessed. Patient-reported outcomes (ThyPRO-39, EQ-5D-5L, neck appearance satisfaction visual analog scale) and clinician-reported scar assessment (Vancouver Scar Scale) will be repeated at Months 1, 3, 6, and 12, with the Voice Handicap Index-10 collected as needed. Laboratory tests (blood count, biochemistry, electrolytes) and immunology samples will be collected every 3 months.

The primary efficacy endpoint is the lymph node volume reduction rate at 12 months after a single IRE ablation. Secondary efficacy endpoints include 12-month lymph node volume reduction rate after single and/or salvage ablation, complete disappearance rate and recurrence rate at 12 months, volume reduction rate at 12 months for lesions located in high-risk anatomical areas, progression-free survival and overall survival, and improvements in quality of life and cosmetic outcomes. Safety endpoints include the incidence of adverse events and serious adverse events graded by NCI CTCAE v5.0, device-related serious adverse events, acute pain tolerability (NRS area under the curve and the proportion of participants with NRS ≥4 of sustained duration), laboratory abnormalities, and changes in voice-related outcomes. Exploratory endpoints include longitudinal changes in immune cell subsets, immune checkpoint and inhibitory molecule expression, and serum cytokine/chemokine profiles. Adverse events will be followed from the last IRE procedure (including salvage ablation) through 12 months.

ELIGIBILITY:
Inclusion Criteria:1: Voluntarily signs a written informed consent form

2: Age ≥ 18 years at the time of enrollment, male or female.

3: ECOG performance status score of 0 or 1.

4: Expected survival time ≥ 12 months.

5: Cervical lymph node metastases confirmed by pathology (core needle biopsy, fine-needle aspiration biopsy, or thyroglobulin testing in fine-needle aspiration washout fluid), and all of the following: ① Thyroid cancer has recurred/metastasized after standard thyroid lobectomy plus lymph node dissection; ② The number of lymph nodes on one side of the neck is ≤ 5, and the maximum long-axis diameter is < 3.0 cm.

6: Not suitable for repeat surgical resection or the patient refuses repeat surgery, or ^131I therapy is ineffective or the patient refuses ^131I therapy.

7: Adequate organ function as defined below: a) Hematologic (no transfusion of blood components or use of hematopoietic growth factors within 7 days prior to initiation of study treatment): i. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (1,500/mm³); ii. Platelet count (PLT) ≥ 100 × 10^9/L (100,000/mm³); iii. Hemoglobin ≥ 90 g/L. b) Renal: i. Calculated creatinine clearance (CrCl)* ≥ 50 mL/min. CrCl (mL/min) is calculated using the Cockcroft-Gault formula: CrCl (mL/min) = {(140 - age) × body weight (kg) × F} / [SCr (mg/dL) × 72] where F = 1 for males and F = 0.85 for females; SCr = serum creatinine. ii. Urine protein ≤ 2+ (dipstick) or 24-hour urine protein < 1.0 g. c) Hepatic: i. Serum total bilirubin (TBil) ≤ 1.5 × ULN (upper limit of normal); for subjects with liver metastases or confirmed/suspected Gilbert's syndrome, TBil ≤ 3 × ULN; ii. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; for subjects with liver metastases, AST and ALT ≤ 5 × ULN. d) Coagulation: International normalized ratio (INR), activated partial thromboplastin time (APTT), and prothrombin time (PT) ≤ 1.5 × ULN. e) Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 50%.

8: Women of childbearing potential must undergo a urine or serum pregnancy test within 3 days prior to the first dose of study treatment (if the urine pregnancy test result cannot be definitively interpreted as negative, a serum pregnancy test must be performed, and the serum result shall prevail), and the result must be negative. If a woman of childbearing potential has sexual intercourse with a male partner who has not been surgically sterilized, she must use an acceptable method of contraception starting from screening and agrees to continue contraception for 180 days after the last dose of the study drug.

9: Male subjects who have not been surgically sterilized and have female partners of childbearing potential must use effective contraception from screening until 180 days after the last dose of the study drug.

10: The subject is willing and able to comply with the visit schedule, treatment regimen, laboratory examinations, and other requirements of the study.

-

Exclusion Criteria:1: History of severe bleeding tendency or coagulation disorders; presence of clinically significant bleeding within 1 month prior to the first ablation treatment, including but not limited to gastrointestinal bleeding, hemoptysis (defined as coughing up or expectorating ≥ 1 teaspoon of fresh blood or small clots, or coughing up blood only without sputum; patients with blood-streaked sputum are allowed to be enrolled), or nasal hemorrhage (excluding minor epistaxis and blood-tinged nasal secretions); continuous anticoagulant therapy within 10 days prior to the first administration of study treatment.

2: History of myocarditis, cardiomyopathy, or malignant arrhythmias. Unstable angina, myocardial infarction, congestive heart failure, or vascular disease (such as an aortic aneurysm at risk of rupture) requiring hospitalization within 12 months prior to the first ablation treatment, or other cardiac damage that may affect the safety evaluation of the study device (e.g., poorly controlled arrhythmias, atrial fibrillation, myocardial ischemia/infarction).

3: Patients who are unable to cooperate with treatment or unable to tolerate general anesthesia.

4: Presence of distant metastases outside the cervical region.

5: Presence of metastatic lymph nodes located in the level VII compartment of the neck.

6: Receipt of ^131I therapy within the past 6 months.

7: Allergy to ultrasound or CT contrast agents, or inability to undergo contrast-enhanced imaging examinations for other reasons.

8: Patients who have undergone neck surgery, local ablation, chemotherapy, or immunotherapy/targeted therapy within the past 3 months.

9: In the opinion of the investigator, ablation needles cannot be safely placed.

10: Presence of metallic implants (plates, screws, etc.) or non-removable implanted catheters in the neck that may affect electric field distribution.

11: Concomitant untreated malignant tumors, or a history of any malignancy within the past 5 years, except for basal cell carcinoma of the skin or carcinoma in situ of the cervix.

12: Concurrent enrollment in another clinical study.

13: Known history of psychiatric disorders, substance abuse, alcoholism, or illicit drug use.

14: Major surgery or severe trauma within 30 days prior to the first ablation treatment, or planned major surgery within 30 days after the first ablation treatment (as determined by the investigator).

15: History within 6 months prior to the first ablation treatment of esophageal or gastric fundal varices, severe peptic ulcer, unhealed wounds, gastrointestinal perforation, enterocutaneous fistula, intestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding; acute exacerbation of chronic obstructive pulmonary disease (COPD) within 1 month prior to the first treatment.

16: Any arterial thromboembolic event, venous thromboembolism of grade ≥ 3 according to CTCAE version 5.0, transient ischemic attack, cerebrovascular accident, hypertensive crisis, or hypertensive encephalopathy within 6 months prior to the first ablation treatment; or current hypertension with systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg despite oral antihypertensive therapy.

17: Any past or current disease, treatment, or laboratory abnormality that may confound the study results, interfere with the subject's full participation in the study, or make participation not in the subject's best interest.

18: Local or systemic diseases not caused by malignant tumors, or tumor-related secondary diseases or symptoms that may lead to high medical risk and/or uncertainty in survival assessment, such as tumor-related leukemoid reaction (white blood cell count > 20 × 10^9/L), manifestations of cachexia (e.g., known weight loss of more than 10% within 3 months prior to screening), etc.

19: Any other condition that, in the opinion of the investigator, makes the subject unsuitable for participation in this study.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Lymph Node Volume Reduction Rate (VRR) at 12 Months） | 12 months after single IRE ablation (Day 0)
  Volume reduction rate (VRR) of the treated target cervical lymph node(s), calculated from imaging-based lymph node volume measurements at baseline and at the 12-month follow-up. Volume will be assessed using contrast-enhanced ultrasound (CEUS).

SECONDARY OUTCOMES:
Lymph Node Volume Reduction Rate (VRR) at 12 Months After Single or Salvage Ablation | 12 months after the last IRE ablation (single ablation on Day 0 or salvage ablation, if performed)
  Volume reduction rate (VRR) of treated target cervical lymph node(s), assessed at 12 months after the last IRE ablation received (single ablation for participants not requiring salvage; salvage ablation for participants receiving salvage). Lymph node volume will be measured by contrast-enhanced ultrasound (CEUS). VRR will be calculated as (baseline volume - follow-up volume) / baseline volume × 100%.
Complete Disappearance Rate of Treated Cervical Lymph Nodes at 12 Months | 12 months after the last IRE ablation (single ablation on Day 0 or salvage ablation, if performed)
  Proportion of treated target cervical lymph node(s) showing complete disappearance at the 12-month follow-up, assessed by contrast-enhanced ultrasound (CEUS). Complete disappearance is defined as no visible target lymph node and no residual enhancement at the treatment site on CEUS. The 12-month assessment will be referenced to the last IRE ablation received (single ablation for participants not requiring salvage; salvage ablation for participants receiving salvage).
Progression-Free Survival (PFS) and Overall Survival (OS) | Up to 24 months after the first IRE ablation (Day 0)
  Time from the first IRE ablation (Day 0) to the first documented disease progression (imaging progression of treated cervical lymph node(s) or new/progressive disease per protocol) or death from any cause, whichever occurs first. Participants without an event will be censored at the date of last contact/follow-up. Disease status will be assessed by scheduled follow-up and confirmed by available clinical records; follow-up contact may include telephone calls.
  Time from the first IRE ablation (Day 0) to death from any cause. Participants alive at the end of follow-up will be censored at the date of last contact/follow-up. Survival status will be obtained through follow-up contact (including telephone follow-up) and available clinical records.
Lymph Node Volume Reduction Rate (VRR) at 12 Months in High-Risk Anatomical Areas (HRA) | 12 months after the last IRE ablation (single ablation on Day 0 or salvage ablation, if performed)
  Volume reduction rate (VRR) of treated target cervical lymph node(s) located in predefined high-risk anatomical areas (HRA), assessed at 12 months after the last IRE ablation received (single ablation for participants not requiring salvage; salvage ablation for participants receiving salvage). Lymph node volume will be measured by contrast-enhanced ultrasound (CEUS). VRR will be calculated as (baseline volume - follow-up volume) / baseline volume × 100%.
Cervical Lymph Node Recurrence Rate at 12 Months | 12 months after the last IRE ablation (single ablation on Day 0 or salvage ablation, if performed)
  Proportion of treated target cervical lymph node(s) with recurrence within 12 months after the last IRE ablation received (single ablation for participants not requiring salvage; salvage ablation for participants receiving salvage). Recurrence is defined as reappearance of the treated lymph node and/or new contrast enhancement at the ablation site on contrast-enhanced ultrasound (CEUS), consistent with viable/recurrent disease per protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- No. 79 Qingchun Road, Shangcheng District, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the primary and secondary outcomes will be shared. This will include participant-level baseline characteristics and eligibility variables; treatment information (IRE procedure details and whether salvage ablation was performed); imaging-derived lymph node measurements/volumes used to calculate volume reduction rate (VRR) and assessments of complete disappearance and recurrence; follow-up dates and event indicators for progression-free survival and overall survival; patient-reported outcomes (ThyPRO-39, EQ-5D-5L, neck appearance satisfaction VAS, and VHI-10 when collected); pain scores (NRS at specified post-procedure time points); adverse event and serious adverse event data (coded and graded per NCI CTCAE v5.0); and laboratory and immune-related variables collected per protocol (e.g., blood counts/biochemistry/electrolytes and de-identified immunology/biomarker measures). A data dictionary and the statistical analysis plan wil
Supporting Information: Study Protocol, SAP, Analytic Code